CLINICAL TRIAL: NCT00538746
Title: Effect of Increased Muscular Work During Different Weaning Strategies in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1500
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2007-10

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Continuous Positive Airway Pressure

ARMS (3):
- 1 (Experimental): BIPAP (Bilevel Positive Airway Pressure) targeted on: TV 6-8 ml/kg, total RR 10-30/min, PEEP and FiO2 regulated on Sat greater than 92% (with spontaneous RR between 20-40%)
  Interventions: Device: BIPAP
- 2 (Experimental): PSV (pressure support ventilation) targeted on: TV 6-8 ml/kg,total RR 10-30/min, PEEP and FiO2 regulated on Sat greater than 92, a minimum of 7 cmH2O of PS is tolerated.
  Interventions: Device: PSV
- 3 (Experimental): PSV+CPAP (continuous positive airway pressure) targeted on: PSV: TV 6-8 ml/kg,total RR 10-30/min, PEEP and FiO2 regulated on Sat greater than 92, a minimum of 7 cmH2O of PS is tolerated, CPAP (5-10 cmH2O) at least 2 hours a day. If during the CPAP periods at least 1 of the criteria T tube test failure occurs, the patients will come back immediately to PSV.
  Interventions: Device: PSV + CPAP

INTERVENTIONS:
Device: BIPAP
  Arms: 1
Device: PSV
  Arms: 2
Device: PSV + CPAP
  Arms: 3

SUMMARY:
Most patients admitted to intensive care units require mechanical ventilation. Weaning from assisted/controlled ventilation begins when we recognize that the patient has recovered adeguately from acute respiratory failure.

If weaning is delayed, costs are increased, as are the risks of nosocomial pneumonia, cardiac-associated morbility, and death. On the other hand, weaning too soon often results in reintubation, which is associated with complications similar to those of prolonged ventilation.

The aim of this trial is to establish an evidence-based approach to weaning and to determine when a patient is ready to be weaned from mechanical ventilation, and what is the best weaning technique.

ELIGIBILITY:
Inclusion Criteria:

1. Age higher than 18 yrs
2. PaO2/FiO2 greater or equal than 150 with PEEP equal or lower than 10, and minute ventilation lower than 15 l/min
3. Temperature lower than 38,5°C
4. Stable hemodynamics: HR 60-125 b/min, SBP 90-160 mmHg without or with dopamine lower than 10 gamma/Kg/min or dobutamine lower than 10 gamma/Kg/min, no acute arrythmias
5. Hb higher than 8 g/dl
6. GCS higher or equal than 9
7. The attending physician has to agree that the patient is in stable conditions and ready to be weaned from the ventilator

Exclusion Criteria:

1. presence of chronic neuromuscular diseases
2. need of surgical intervention within the next 72 hours
3. difficult tracheal intubation
4. tracheostomized patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-02

PRIMARY OUTCOMES:
1. Days of intubation 2. Days of mechanical ventilation | 28 days

SECONDARY OUTCOMES:
1. The day of eventual tracheostomy 2. Organ Failure 3. The mortality at 28° day 4. Outcome at 6 months | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pelosi, Professor, Principal Investigator — Universita' degli Studi dell'Insubria
Locations (1):
- Ospedale di Circolo e Fondazione Macchi, Varese, Varese, Italy